CLINICAL TRIAL: NCT07055958
Title: Effect of Metformin as Add-on Therapy in Levodopa Treated Parkinson's Disease Patients: Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Effect of Metformin as Add-on Therapy in Levodopa Treated Parkinson's Disease Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, RUKHSANA AKTER, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5246
Record Dates: First submitted 2025-05-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Metformin, Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin- Patients receiving Levodopa with Metformin (Experimental): Dosage form- Tab. Metformin 500 mg, Frequency - once daily, Duration - 8 weeks
  Interventions: Drug: Metformin
- Control - Patients receiving Levodopa with Placebo (Placebo Comparator): placebo of Tab. Metformin 500 mg, frequency- once daily, duration- 8 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Metformin — Metformin's chemical name is 1,1-Dimethylbiguanide, a molecular formula of C4H11N5. Beyond its well established antihyperglycemic impact, metformin demonstrated anti-oxidant and anti-inflammatory activities contributing its potential benefits in conditions associated with inflammation and oxidative stress. Furthermore, metformin rapidly crosses the blood brain barrier and disperses into several brain regions presenting an ideal therapeutic option for the treatment of PD.
  Arms: Metformin- Patients receiving Levodopa with Metformin
Other: placebo — placebo of tab. Metformin of same shape
  Arms: Control - Patients receiving Levodopa with Placebo

SUMMARY:
The goal of this clinical trial is to learn that metformin has effect on motor aspects of daily living and oxidative stress in levodopa treated Parkinson disease patients. Researcher will compare drug metformin to a placebo. Participants will take metformin or placebo for 8 weeks.

DETAILED DESCRIPTION:
This clinical trial is an effort to explore whether administration of metformin has effect on motor aspects of daily living and oxidative stress in levodopa treated Parkinson's disease patients. After completion of necessary formalities, each participant will be assessed by translated and validated Bangla version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part questionnaire and malondialdehyde (MDA) and glutathione (GSH) will be measured at baseline and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed mild to moderate PD patients taking Levodopa
* Age 18 years and older
* Sex : Any

Exclusion Criteria:

* Secondary causes of Parkinsonism
* Prior stereotactic surgery for PD
* Suffering from active malignancy
* Known hypersensitivity to metformin
* Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
motor aspects of daily living | 8 weeks
  motor aspects of daily living in MDS-UPDRS rating scale (Movement Disorder Society- sponsored revision of the Unified Parkinson's Disease Rating Scale). The score of Part 2 of this scale i.e. motor experiences of daily living is 13.

SECONDARY OUTCOMES:
1. Plasma Malondealdehyde (MDA) level in micromole/litre. 2. Erythrocyte Glutathione (GSH) level in mg/ml. | 8 weeks
  Malondealdehyde is oxidative stress marker. Glutathione is anti-oxidant.
1. Erythrocyte glutathione level in mg/ml 2. Erythrocyte Glutathione (GSH) level in mg/ml. | 8 weeks
  Glutathione is an anti-oxidant Glutathione is anti-oxidant.
Comparison of adverse effects in percentage | 8 weeks
  Adverse effects in Metformin treated and placebo treated patients

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh